CLINICAL TRIAL: NCT03417700
Title: Vitamin D as a Factor Modifying Adaptation to Diverse Forms of Exercise
Brief Title: Vitamin D as a Factor Modifying Adaptation to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Principal Investigator, Robert Olek, Associate Professor, Gdansk University of Physical Education and Sport
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/15/B/NZ7/00976
Record Dates: First submitted 2017-11-30; First posted 2018-01-31 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Vitamin D3 Deficiency
Keywords: vitamin D; exercise; training; aging
MeSH Terms: conditions — Motor Activity | interventions — Vitamin D; Control Groups; Resistance Training

STUDY DESIGN:
Intervention Model Description: Model I
  Women and men over 65 years old will participate in the training programme. All subjects will undergo a medical check-up before being subject to exercise. All procedures will be performed with the approval from the Bioethical Committee of the Regional Medical Society in Gdansk. One week prior to the beginning of the experiment, a battery of physiological and psychological tests will be performed. The same procedure will be repeated after the training period.
  In addtition to training, supplementation of vitamin D (800IU and 4000IU) will be administered.
  Model II
  Young women will participate in the training programme. They will perform a high-intensity circuit training according to the ACSM. They will perform a single session of HICT and 12 units of HICT regularly. One week prior to the beginning of the experiment, a battery of physiological and psychological test will be performed. The same procedure will be repeated after the training period.
Who Masked: Investigator
Masking Description: Participants will receive vitamin D supplementation, but the dose will be known only to one investigator, who will be not be participating in any other assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training NW (Experimental): exercise and supplementation
  Interventions: Dietary Supplement: NW training; Dietary Supplement: Placebo
- Training HICT and vitamin D (Experimental): Training HICT plus vitamin D
  Interventions: Dietary Supplement: NW training; Dietary Supplement: Placebo; Dietary Supplement: HICT
- Placebo (Experimental): placebo Vitamin D
  Interventions: Dietary Supplement: NW training

INTERVENTIONS:
Dietary Supplement: NW training — NW training
  Other Names: Training; vitamin D
Dietary Supplement: Placebo — training with placebo
  Other Names: Control group
  Arms: Training HICT and vitamin D; Training NW
Dietary Supplement: HICT — Training and vitamin D
  Other Names: resistance training
  Arms: Training HICT and vitamin D

SUMMARY:
Physical activity is a recommended, indispensable element of a healthy lifestyle as well as a countermeasure against many diseases often accompanied by the acute or chronic low grade inflammation. Papers published in recent years have demonstrated the anti-inflammatory effect of exercise. Based on current knowledge of the topic, own experience and preliminary work, it is expected the proposed research to provide information on the mechanism either determining or limiting pro-healthy effects of exercise in different age groups of people. Three different training programmes will be investigated. Specific goals of the project include the following:

1. Establish, whether regular Nordic Walking training and HIIT can reduce the low-grade systemic inflammation and which type of training is the most effective at doing so.
2. Establish, whether regular training can prevent muscle sarcopenia and assess if those changes are related to the concentration of the autophagy-inducing stress protein, HMGB1.
3. Establish, whether regular Nordic Walking training alters iron metabolism and evaluate its correlation with the inflammatory markers and bone-morphogenesis.
4. Establish, whether muscle-released irisin signals growth in the BDNF concentration in response to exercise and if these changes improve cognitive function.
5. Establish, whether Nordic Walking or HIIT training effectively improve the blood lipid profile and aerobic capacity, and if these effects correlate with the blood 25-OHD concentration.
6. Establish, whether concentration of vitamin D alters adaptation to training and modifies immunological response to regular training process.

DETAILED DESCRIPTION:
The mechanism behind the anti-inflammatory effect of exercise is not fully understood. In some cases physical activity has proven almost/completely ineffective in reducing systemic inflammation. Thus, evaluating factors, which modify this response, is of particular significance. One of them may be related to iron metabolism. It is has been suggested that regular training reduces body iron stores, which can contribute to the anti-inflammatory response. Consequently, one of the anti-inflammatory effects of exercise can be related to changes in iron metabolism. Nevertheless, our preliminary data demonstrated that eight months of Nordic Walking training did not reduce body iron stores in approx. 25% of subjects, even if some of them were characterized by high blood ferritin (good indicator of body iron stores). This may be related to the effect of exercise on the concentration of hepcidin (main regulator of iron absorption, which acts as a negative regulator of iron efflux). It is well documented that a single bout of exercise induces an increase in blood hepcidin; however, data on the effect of regular training on the hepcidin concentration are limited.

Vitamin D is another factor, which could influence the anti-inflammatory effect of exercise. It has been suggested that individuals involved in physical activity have higher concentrations of 25OHD (indicator of vitamin D status). Vitamin D inhibits the expression of pro-inflammatory cytokines, which is considered the main mechanism of its anti-inflammatory action. It is worth noting that population in Poland is characterized by low status of vitamin D. Thus, it is possible that the anti-inflammatory effect of exercise will be modified by the vitamin status. Moreover, vitamin D has been shown to protect against muscle atrophy both in elderly and younger people. Its concentration has been correlated with muscle strength.

Inflammation has been observed to be associated with an increase of the autophagy-inducing stress protein, HMGB1, which mediates muscle atrophy. Measurement of plasma amino acid profile will be helpful to assess the impact of exercise on muscle proteolysis. Moreover, the link between exercise, vitamin D status and HMGB1 has not yet been established. In addition, a range of interactions induced by exercise involves the release of the newly discovered protein, irisin, form the muscle and its improving effect on the cognitive function through the synthesis of brain-derived neurotrophic factor (BDNF). Data on the effect of regular training on irisin concentration in elderly people is lacking.

Overall, our research interest focuses on the role of the factors mediating the anti-inflammatory effect of exercise and the way they stimulate or inhibit adaptive changes. The proposed project draws on our long experience in investigating the effects of exercise on iron metabolism as well as other physical methods supporting the anti-inflammatory action of physical activity. Latest published papers indicate that the concentration of vitamin D, also in training adaptation, can modulate immunological response to exercise. Therefore, verifying our hypothesis would also allow us to determine if the concentration of vitamin D can limit adaptation to physical activity.

ELIGIBILITY:
Inclusion Criteria:

no illness medical check

Exclusion Criteria:

uncontrolled hypertension (diastolic blood pressure over 100 mmHg), a history of cardiac arrhythmia, cardio-respiratory disorders, advanced osteoporosis, clinical diagnosis of Alzheimer's Disease

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
The influence of vitamin D on physical performance in aging people | Values at baseline will be compared to values recorded 12 weeks and 3 months after the training programme.
  To verify if training supported by vitamin D supplementation will bring better effects

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Ziemann, Principal Investigator — Gdansk University of Physical Education and Sport, Poland
Locations (2):
- Poland (2):
  - University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship
  - Ziemann Ewa, Sopot, Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: No
Written-up results of research will be submitted for publication to international journals.

REFERENCES:
- [Result] Gmiat A, Mieszkowski J, Prusik K, Prusik K, Kortas J, Kochanowicz A, Radulska A, Lipinski M, Tomczyk M, Jaworska J, Antosiewicz J, Ziemann E. Changes in pro-inflammatory markers and leucine concentrations in response to Nordic Walking training combined with vitamin D supplementation in elderly women. Biogerontology. 2017 Aug;18(4):535-548. doi: 10.1007/s10522-017-9694-8. Epub 2017 Mar 18. PMID 28316011
- [Result] Prusik K, Kortas J, Prusik K, Mieszkowski J, Jaworska J, Skrobot W, Lipinski M, Ziemann E, Antosiewicz J. Nordic Walking Training Causes a Decrease in Blood Cholesterol in Elderly Women Supplemented with Vitamin D. Front Endocrinol (Lausanne). 2018 Feb 20;9:42. doi: 10.3389/fendo.2018.00042. eCollection 2018. PMID 29515518
- [Result] Walentukiewicz A, Lysak-Radomska A, Jaworska J, Prusik K, Prusik K, Kortas JA, Lipinski M, Babinska A, Antosiewicz J, Ziemann E. Vitamin D Supplementation and Nordic Walking Training Decreases Serum Homocysteine and Ferritin in Elderly Women. Int J Environ Res Public Health. 2018 Sep 20;15(10):2064. doi: 10.3390/ijerph15102064. PMID 30241318
- [Result] Mieszkowski J, Niespodzinski B, Kochanowicz A, Gmiat A, Prusik K, Prusik K, Kortas J, Ziemann E, Antosiewicz J. The Effect of Nordic Walking Training Combined with Vitamin D Supplementation on Postural Control and Muscle Strength in Elderly People-A Randomized Controlled Trial. Int J Environ Res Public Health. 2018 Sep 7;15(9):1951. doi: 10.3390/ijerph15091951. PMID 30205445
- [Result] Gmiat A, Jaworska J, Micielska K, Kortas J, Prusik K, Prusik K, Lipowski M, Radulska A, Szupryczynska N, Antosiewicz J, Ziemann E. Improvement of cognitive functions in response to a regular Nordic walking training in elderly women - A change dependent on the training experience. Exp Gerontol. 2018 Apr;104:105-112. doi: 10.1016/j.exger.2018.02.006. Epub 2018 Feb 9. PMID 29432893
- [Result] Kortas J, Kuchta A, Prusik K, Prusik K, Ziemann E, Labudda S, Cwiklinska A, Wieczorek E, Jankowski M, Antosiewicz J. Nordic walking training attenuation of oxidative stress in association with a drop in body iron stores in elderly women. Biogerontology. 2017 Aug;18(4):517-524. doi: 10.1007/s10522-017-9681-0. Epub 2017 Feb 22. PMID 28229255